CLINICAL TRIAL: NCT00216762
Title: Phase I/II Open Label Evaluation of the Safety and Efficacy of Rituximab in Patients With Chronic Urticaria (The Rituximab Urticaria Study - "RUSTY")
Brief Title: Safety Study of Rituximab (Rituxan®) in Chronic Urticaria
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Full Clinical Hold
Sponsor: Johns Hopkins University (Other)
Collaborators: Genentech, Inc. (Industry)
Responsible Party: Principal Investigator, Clifton O Bingham, Principal Investigator, Johns Hopkins University
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NA_00000857
Record Dates: First submitted 2005-09-16; First posted 2005-09-22 (Estimated); Last update posted 2015-09-02 (Estimated); Status verified 2015-08

CONDITIONS: Urticaria
Keywords: Urticaria; Hives
MeSH Terms: conditions — Urticaria | interventions — Rituximab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: Rituximab — Rituxan ® 1000 mg IV x 2 infusions, 2 weeks apart
  Other Names: Rituxan ®

SUMMARY:
This study is being done to find out if a drug called Rituxan (Rituximab) is safe and effective in treating people with chronic urticaria (hives) with persistent symptoms in spite of taking antihistamines.

DETAILED DESCRIPTION:
Rituximab (Rituxan®) is a recombinant chimeric monoclonal antibody that binds to a molecule (CD20) that is present on the surface of B lymphocytes. The product is approved for the treatment of non-Hodgkin's lymphoma and has been investigated for the treatment of a number of autoimmune diseases including rheumatoid arthritis (Edwards 2004) and lupus (Looney 2004, Leandro 2002). As in most rheumatoid arthritis studies, the medication will be administered in this study as a series of two intravenous infusions given 2 weeks apart.

Many cases of chronic urticaria (hives) are though to be driven by an autoimmune mechanism (Kaplan 2002, Grattan 2002). It is our hypothesis that by interfering with the autoimmune process, potentially by decreasing the levels of autoantibodies or by interfering with other mechanisms that cause basophil and mast cell activation, improvments in signs and symptoms will be seen.

Given the effectiveness demonstrated for Rituximab in other autoimmune conditions, we will conduct a pilot open label investigation of 15 patients with chronic urticaria to determine the safety and effectiveness of Rituximab in this disease. All patients will receive the medication; there will be no placebo group in this study. Rituximab is not currently indicated for the treatment of this condition however.

We will evaluate the safety of the Rituximab in 15 patients with urticaria as well as studies of antibody levels and cellular function. We will also evaluate clinical outcomes such as itch score, sleep disturbance, and quality of life. After receivng the Rituximab treatment, we will begin to taper antihistamines and other medications used to control urticaria symptoms.

ELIGIBILITY:
Major Inclusion Criteria:

* Chronic urticaria defined as symptoms >50% of the days or 3 days per week for more than 12 weeks
* Previous requirement for sustained or recurrent use of corticosteroids OR requirement for immunomodulatory treatment for urticaria (eg hydroxychloroquine, sulfasalazine, dapsone, cyclosporine, IVIg, etc) OR ongoing symptoms for at least 6 months duration with failure to respond at least maximally approved dosages of 2 different antihistamine therapies
* Chronic therapy with stable doses of antihistamines for at least 4 weeks. Patients may be taking more than one antihistamine or be taking combinations of antihistamines and leukotriene receptor antagonists
* High baseline score for pruritis (at least 2 on a 3 point scale)
* No underlying etiology clearly defined for urticaria
* Evidence of underlying autoimmunity as evidenced by clinical and laboratory criteria
* Concomitant use of hydroxychloroquine, sulfasalazine, or dapsone permitted if doses stable for at least 12 weeks
* Negative serum pregnancy test (for women of child-bearing age)
* Men and women of reproductive potential must agree to use an acceptable method of birth control during treatment and for twelve months (1 year) after completion of treatment.
* No planned elective surgical procedures for at least 6 months

Major Exclusion Criteria:

* Concomitant use of corticosteroids
* Current use of immunosuppressive medication (cyclosporine, IVIg, methotrexate, cyclophosphamide). Any such medication will be discontinued for at least 6 weeks before screening.
* Treatment with any investigational agent within 4 weeks of screening or 5 half-lives of the investigational drug (whichever is longer)
* Receipt of a live vaccine within 4 weeks prior to randomization
* Previous treatment with Rituximab (MabThera® / Rituxan®)
* Prior antibody therapy
* History of severe allergic or anaphylactic reactions to humanized or murine monoclonal antibodies
* Known history of HIV seropositivity (testing will be performed at screening)
* History of Hepatitis B and/or Hepatitis C (Hep BsAg and Hep C Ab will be obtained at screening)
* History of recurrent significant infection or history of recurrent bacterial infections
* Known active bacterial, viral, fungal, mycobacterial, or other infection (including tuberculosis or atypical mycobacterial disease, but excluding fungal infections of nail beds)
* Any major episode of infection requiring hospitalization or treatment with i.v. antibiotics within 4 weeks of screening or oral antibiotics within 2 weeks prior to screening
* Known immunodeficiency syndrome, hypogammaglobulinemia, etc.
* Systemic lupus erythematosus
* Pregnancy (a negative serum pregnancy test will be performed for all women of childbearing potential within 7 days of treatment) or lactation
* Malignancies within the last five years, with the exception of adequately treated basal or squamous cell carcinoma of the skin or carcinoma in situ of the cervix.
* Atopic dermatitis
* Clinically relevant medical conditions (cardiovascular including poorly controlled hypertension or coronary artery disease, pulmonary, metabolic, renal, hepatic, psychiatric) or clinical laboratory finding giving reasonable suspicion of a disease or condition that contraindicates the use of an investigational drug or that may affect the interpretation of the results or render the patient at high risk from treatment complications
* Plans or need to receive live viral vaccination over course of the study (e.g. Flu-Mist TM)

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2006-01; Primary Completion 2007-05 (Actual); Study Completion 2007-05 (Actual)

PRIMARY OUTCOMES:
Safety of Rituximab infusions in this patient population | 1 year or time until reconstitution of B cells

CONTACTS AND LOCATIONS:
Overall Officials: Clifton O. Bingham, III, MD, Principal Investigator — Johns Hopkins University, Divisions of Rheumatology and Allergy and Clinical Immunology
Locations (1):
- Johns Hopkins University, Bayview Medical Center, Baltimore, Maryland, United States

REFERENCES:
- [Background] Kaplan AP. Clinical practice. Chronic urticaria and angioedema. N Engl J Med. 2002 Jan 17;346(3):175-9. doi: 10.1056/NEJMcp011186. No abstract available. PMID 11796852
- [Background] Grattan CE, Sabroe RA, Greaves MW. Chronic urticaria. J Am Acad Dermatol. 2002 May;46(5):645-57; quiz 657-60. doi: 10.1067/mjd.2002.122759. PMID 12004303
- [Result] Looney RJ, Anolik JH, Campbell D, Felgar RE, Young F, Arend LJ, Sloand JA, Rosenblatt J, Sanz I. B cell depletion as a novel treatment for systemic lupus erythematosus: a phase I/II dose-escalation trial of rituximab. Arthritis Rheum. 2004 Aug;50(8):2580-9. doi: 10.1002/art.20430. PMID 15334472
- [Result] Edwards JC, Szczepanski L, Szechinski J, Filipowicz-Sosnowska A, Emery P, Close DR, Stevens RM, Shaw T. Efficacy of B-cell-targeted therapy with rituximab in patients with rheumatoid arthritis. N Engl J Med. 2004 Jun 17;350(25):2572-81. doi: 10.1056/NEJMoa032534. PMID 15201414
- [Result] Leandro MJ, Edwards JC, Cambridge G, Ehrenstein MR, Isenberg DA. An open study of B lymphocyte depletion in systemic lupus erythematosus. Arthritis Rheum. 2002 Oct;46(10):2673-7. doi: 10.1002/art.10541. PMID 12384926